CLINICAL TRIAL: NCT00868153
Title: Levonorgestrel Releasing Intrauterine Device (Mirena) in Idiopathic Menorrhagia
Brief Title: Mirena in Idiopathic Menorrhagia
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14494; MA0501
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Idiopathic Menorrhagia
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Levonorgestrel IUS (Mirena , BAY86-5028)

INTERVENTIONS:
Drug: Levonorgestrel IUS (Mirena , BAY86-5028) — One group

SUMMARY:
This is an open-label, uncontrolled, multi-centre observational study that analyses a follow-up of 1600 women with dysfunctional uterine bleeding (idiopathic menorrhagia) over a period of one year.The patients evaluated at four visits, beginning with the insertion visit and 3, 6 and 12 months after insertion.

ELIGIBILITY:
Inclusion Criteria:

* Woman diagnosed with idiopathic Menorrhagia according to assessment of the investigator and according to international guidelines. These woman should also accept to be on contraception during the time period that they have Mirena in situ.
* Age limit 30-45
* BMI= 18-34
* Signed informed consent

Exclusion Criteria:

* Medical conditions featured in the Mirena data sheet (See Appendix 1) that contraindicate its use, listed below:
* Known or suspected pregnancy; current or recurrent pelvic inflammatory disease; infection of the lower genital tract; postpartum endometritis; septic abortion during the past three months; cervicitis; cervical dysplasia; uterine or cervical malignancy; undiagnosed abnormal uterine bleeding; congenital or acquired abnormality of the uterus including fibroids if they distort the uterine cavity; conditions associated with increased susceptibility to infections; acute liver disease or liver tumor; known hypersensitivity to any of the constituents of the product.
* Nulliparity
* Consumption of Iron, Antiprostaglandins, hormonal drugs and any medication that could effect bleeding should be stopped at least 3 months before the first visit and should not be used during the course of the study.
* History of diabetes mellitus,cardiovascular disease and thyroid abnormalities
* Anticoagulation therapy
* Cancer history including breast cancer.

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women diagnosed with idiopathic menorrhagia, age 30-45, BMI 18-34
Sampling Method: Non-Probability Sample
Enrollment: 1125 (Actual)
Dates: Start 2004-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the improvement in the quality of life and the degree of satisfaction of women with idiopathic menorrhagia treated with Mirena | At vist 1 and 4

SECONDARY OUTCOMES:
Information about the pattern of menstrual bleeding recorded in an ongoing way throughout the duration of the study | Every visit
The health-related quality of life questionnaire SF-36 at Visits 1 and 4 | Visit 1 and 4
The user satisfaction as recorded at Visit 4 | visit 4
Adverse reactions recorded in an ongoing way throughout the duration of the study | every visit
Laboratory parameters as measured at Visits 1 and 4 | visit 1 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- Many Locations, Bulgaria
- Many Locations, Croatia
- Many Locations, India
- Many Locations, Jordan
- Many Locations, Kuwait
- Many Locations, Pakistan
- Many Locations, Romania
- Many Locations, Russia
- Many Locations, Saudi Arabia
- Many Locations, Serbia
- Many Locations, Sri Lanka
- Many Locations, Turkey (Türkiye)
- Many Locations, United Arab Emirates